CLINICAL TRIAL: NCT04918888
Title: SARS-CoV-2 Vaccination in Oncologic Patients: A Prospective, Explorative Study
Brief Title: COVID-19 Vaccination in Oncologic Patients
Acronym: VINCI
Status: Completed | Type: Observational
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Other Study IDs: ECS 1048/2021
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Covid19; Oncologic Disorders
Keywords: radiotherapy; SARS-CoV-2 vaccine; immune response; oncologic therapies; immunosuppression; SARS-CoV-2 S binding antibodies; vaccination willingness; vaccination side effects
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Overall study population: All new oncologic patients of the outpatient-clinic of the department of radiooncology
- First dose received (Subpopulation 1): Patients, who received one or two doses of SARS-CoV-2 vaccine prior to radiotherapy
- Vaccination during therapy (Subpopulation 2): Patients, who will receive at least one dose of SARS-CoV-2 vaccine during or up to 6 weeks after radiotherapy

SUMMARY:
Evaluating the vaccination willingness in oncologic patients over six months as well as estimating the effects of radiotherapy/systemic anticancer treatment on the efficacy and toxicity of currently approved SARS-CoV-2 vaccines

DETAILED DESCRIPTION:
All patients that present themselves newly at the outpatient-clinic of the Department of Radiooncology at the Ordensklinikum Linz GmbH, Barmherzige Schwestern during a period of six months are eligible for participation. After being informed about the study, the participants answer a short structured interview regarding vaccination status and vaccination willingness. Patients who already received one or two doses of SARS-CoV-2 vaccine are eligible for the study's subpopulation 1, with the main focus of quantifying SARS-CoV-2 S binding antibody titres after at least 35 days from initial vaccination. Patients who are to receive at least one dose of vaccine during or up to six weeks after radiotherapy are eligible for subpopulation 2, comprising serial measurements of SARS-CoV-2 S binding antibody titres before and after vaccination.

ELIGIBILITY:
Inclusion Criteria:

Study population for the cross-sectional study (patients with previous SARS-CoV-2 infection of previous vaccination, evaluation of willingness to get vaccinated:

* Patients with solid tumors/haematooncologic diseases regardless of stage that seek treatment in the outpatient clinic of the department of radiooncology from April to September 2021 who will undergo active treatment.
* Age: 18-120 years Patients that undergo radiotherapy, radio-chemotherapy, radio-hormonotherapy or radio-immunotherapy during the investigation period.

Longitudinal study:

* Patients that have not yet received SARS-CoV-2 vaccination, but are scheduled to get the first dose during or up to six weeks after active therapy.
* Age: 18-120 years

Exclusion Criteria:

* Lack of written consent
* Patients, that are mentally or physically incapable of completing a questionnaire
* Age: < 18 years
* A previous SARS-CoV-2 infection is no exclusion criteria!

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: new patients of the department for radiooncology at the Ordensklinikum Barmherzige Schwestern Linz
Sampling Method: Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Quantification of vaccination willingness | once directly after enrollment
  guided interview

SECONDARY OUTCOMES:
SARS-CoV-2 antibody titre in already vaccinated patients | >= 35 days post first dose
SARS-CoV-2 antibody titre in patients vaccinated during antineoplastic treatment | baseline and 7, 14,21,28,35, 182 and 365 days post first dose
  Development of antibody titre in patients who received the first or second dose of SARS-CoV-2 vaccine during radiotherapy, Longitudinal quantification of binding antibodies
Qualitive assessment of reasons to reject vaccination | once directly after enrollment
  guided interview
Qualitive assessment of comorbidities | once after enrollment prior to vaccination
  (in respect of the gravity of a SARS-CoV-2 infection corresponding to the WHO-grading), guided interview
Kind and dosage of accompanying systemic therapies | once after enrollment
Modalities and duration of the radiotherapy (irradiated region, single dose overall dose) | once after enrollment
Previous SARS-CoV-2 infection (Rate of undetected cases via antibody detection, for known previous disease: evaluation of severity) | once directly after enrollment and ev. at >= 35 days after first dose
  guided interview, conducted again at day 35 after the first dose for patients who receive radiotherapy during the first dose of vaccination
Qualitative and quantitative assessment of local/systemic side effects of the SARS-CoV-2 vaccination | 35 days after vaccination
  questionnaire
incidence of a symptomatic SARS-CoV-2 infection (duration, extent and severity) | 35 days after vaccination
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hans Geinitz, Univ.-Prof., Principal Investigator — Ordensklinikum Linz GmbH, Barmherzige Schwestern
Locations (2):
- Austria (2):
  - Department of Radiooncology, Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz, Upper Austria
  - Ordensklinikum Linz GmbH, Barmherzige Schwestern, Linz, Upper Austria

REFERENCES:
- [Derived] Geinitz H, Silberberger E, Spiegl K, Feichtinger J, Wagner H, Hermann P, Brautigam E, Track C, Weis EM, Venhoda C, Huppert R, Spindelbalker-Renner B, Zauner-Babor G, Nyiri DV, Karasek N, Erdei M, Gheju R, Gruber G, Egger M, Dieplinger B. SARS-CoV-2 vaccination willingness and humoral vaccination response in radiation oncology patients. Vaccine. 2024 Feb 6;42(4):945-959. doi: 10.1016/j.vaccine.2024.01.006. Epub 2024 Jan 20. PMID 38246842